CLINICAL TRIAL: NCT00118209
Title: Phase III Randomized Study of R-CHOP V. Dose-Adjusted EPOCH-R With Molecular Profiling in Untreated De Novo Diffuse Large B-Cell Lymphomas
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50303; CDR0000433265 (Other: NCI Physician Data Query); NCI-2009-00480 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA031946 (NIH); U10CA180821 (NIH); NCT00234351 (obsolete NCT alias)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2020-04-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Large B Cell Lymphoma
MeSH Terms: interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Etoposide; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - R-CHOP (Active Comparator): Patients receive the following treatment:
  * Rituximab 375 mg/m^2 IV infusion on Day 1 prior to CHOP chemotherapy
  * Cyclophosphamide 750 mg/m^2 IV on Day 1
  * Doxorubicin 50 mg/m^2 IV on Day 1
  * Vincristine 1.4 mg/m^2 IV (2 mg cap) on Day 1
  * Prednisone 40 mg/m^2/day PO on Days 1-5
  * filgrastim or pegfilgrastim as defined in the protocol
  Required ancillary medications is administered during all cycles as defined in the protocol.
  Cycles will be repeated every 21 days for 6 treatment cycles. Restaging will occur after Cycles 4 and 6.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone; Drug: filgrastim; Drug: pegfilgrastim
- Arm B - DA-EPOCH-R (Experimental): Patients receive the following treatment:
  Cycle 1 Doses:
  * Rituximab 375 mg/m^2 IV infusion on Day 1 prior to EPOCH chemotherapy
  * Doxorubicin 10 mg/m^2/day CIVI on Days 1-4
  * Etoposide 50 mg/m^2/day CIVI on Days 1-4
  * Vincristine 0.4 mg/m^2/day (no cap) CIVI on Days 1-4 (total 1.6 mg/m2 over 96 hours)
  * Cyclophosphamide 750 mg/m^2 IV on Day 5 (following completion of 96 hour infusions)
  * Prednisone 60 mg/m^2 PO BID on Days 1-5
  * Administer filgrastim 480 mcg subcutaneous daily from Day 6 until ANC > 5000 after the nadir (nadir usually between Days 10-12) or for 10 days (Days 6-15) if the ANC is not being monitored, during every cycle.
  Doses for subsequent cycles will be determined by the absolute neutrophil (ANC) or platelet nadir from the previous cycle.
  Required ancillary medications are administered during all cycles as defined in the protocol.
  Cycles will be repeated every 21 days for a maximum of 6 cycles. Restaging will occur after Cycles 4 and 6.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone; Drug: etoposide; Drug: filgrastim

INTERVENTIONS:
Biological: rituximab — IV
Drug: cyclophosphamide — IV
Drug: doxorubicin — IV or CIVI
Drug: vincristine — IV or CIVI
Drug: prednisone — oral
Drug: etoposide — CIVI
  Arms: Arm B - DA-EPOCH-R
Drug: filgrastim — IV
Drug: pegfilgrastim — IV
  Arms: Arm A - R-CHOP

SUMMARY:
This randomized phase III trial studies rituximab when given together with two different combination chemotherapy regimens to compare how well they work in treating patients with diffuse large B-cell non-Hodgkin's lymphoma. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving rituximab together with combination chemotherapy may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective when given with rituximab in treating diffuse large B-cell non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying rituximab when given together with two different combination chemotherapy regimens to compare how well they work in treating patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the event-free survival of rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, prednisone (R-CHOP) versus dose-adjusted (DA-) etoposide, prednisone, vincristine sulfate, doxorubicin hydrochloride, cyclophosphamide, and rituximab (EPOCH-R) chemotherapy in untreated cluster of differentiation (CD)20 positive (+) diffuse large B-cell lymphomas.

II. To develop a molecular predictor of outcome of R-CHOP and DA-EPOCH-R chemotherapy using molecular profiling.

SECONDARY OBJECTIVES:

I. To compare the response rates, overall survival and toxicity of R-CHOP versus DA-EPOCH-R.

II. To define the pharmacogenomics of untreated diffuse large B-cell lymphoma (DLBCL) and correlate clinical parameters (toxicity, response, survival outcomes and laboratory results) with molecular profiling.

III. To assess the use of molecular profiling for pathological diagnosis. IV. To identify new therapeutic targets using molecular profiling. V. To perform a comprehensive analysis of somatic alterations to the tumor genome and to understand which genomic alterations are somatically acquired by the tumor and which are encoded in the germ line of the patient.

VI. To identify biomarkers of response to chemotherapy by fludeoxyglucose F 18 (FDG)-positron emission tomography (PET)/computed tomography (CT) imaging that are predictive of histopathologic remissions and survival in patients with stage I (mediastinal), II, III, or IV untreated DLBCL.

VII. To evaluate the use of semiquantitative measurements of FDG uptake in defining FDG-PET/CT based biomarkers of response to chemotherapy in patients with DLBCL.

VIII. To determine whether FDG-PET/CT measurements of tumor response after the second cycle of chemotherapy can predict clinical response.

IX. To establish a standardized protocol for FDG-PET/CT image acquisition. X. To determine additional FDG-PET/CT parameters (e.g., the ratio of tumor maximum standard uptake value [SUVmax] to liver SUVmean; SUVs corrected for body surface area and lean body mass; nuclear medicine physician's assessment) and evaluate their utility in refining FDG-PET/CT based biomarkers of response to therapy.

XI. To evaluate inter-institutional reproducibility of FDG-PET/CT measurements for this indication.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ELIGIBILITY:
1. Histologically documented de novo CD20+ DLBCL with stage II, III or IV disease.

   * Stage I primary mediastinal (thymic) DLBCL is also eligible.
   * Patients with an underlying low-grade lymphoma, such as a transformed lymphoma or low-grade lymphoma in the bone marrow, are not eligible.
   * Diagnosis should be based on an adequate tissue sample, including open biopsy or core needle biopsy.
   * Needle aspiration for primary diagnosis is unacceptable.
   * Patients must have one of the following WHO classification subtypes:

     * Diffuse large B-cell lymphoma (includes morphological variants: centroblastic, immunoblastic, T-cell/histiocyte rich, and anaplastic)
     * Mediastinal (thymic) large B-cell lymphoma
     * Intravascular large B-cell lymphoma
   * Note: Failure to submit a pathology block within 60 days of patient registration will be considered a major protocol violation.

     * Fresh (frozen) tumor biopsy must be available or attempted. A frozen tumor biopsy equivalent to a minimum of four at least 16 gauge needle cores is an important component of this study.
     * Patients without adequate frozen material should have a biopsy performed to obtain material.
     * If a biopsy is performed and does not yield adequate material, the patient is still eligible for the study. If a biopsy cannot be done safely, the patient may still be eligible for the study if permission is granted.
   * Note: This study does not allow concurrent radiation unless a patient has a documented CNS treatment failure with no systemic failure.
2. No prior cytotoxic chemotherapy or rituximab. Patients may be entered if they have received prior limited field radiation therapy or a short course of glucocorticoids (< 10 days) for an urgent local disease complication at diagnosis (e.g., cord compression, SVC syndrome). Patients who have received chemotherapy for prior malignancies are not eligible.
3. Age ≥ 18 years
4. ECOG Performance Status 0-2
5. No active ischemic heart disease or congestive heart failure. If there is suspicion of cardiac disease, a cardiac ejection fraction must show LVEF > 45%, but the study is not required
6. No known lymphomatous involvement of the CNS. A lumbar puncture prior to study is not required in the absence of neurological symptoms
7. No known HIV disease. Patients with a history of intravenous drug abuse or any other behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus. Patients who test positive or who are known to be infected are not eligible.
8. Non pregnant and non-nursing. Treatment would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective form of contraception.
9. Patients with active medical processes (e.g., uncontrolled bacterial or viral infection, bleeding) not related to their lymphoma should be excluded.
10. Required Initial Laboratory Values (unless non-Hodgkin lymphoma):

    * ANC ≥ 1000/μL
    * Platelets ≥ 100,000/μL
    * Creatinine≤ 1.5 mg/dL or creatinine clearance ≥ 50 cc/min
    * Total Bilirubin ≤ 2 mg/dL (unless a history of Gilbert's Disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wyndham H. Wilson, MD, PhD, Study Chair — National Cancer Institute (NCI); Andrew D. Zelenetz, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (47):
- United States (47):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Naval Medical Center - San Diego, San Diego, California
  - Saint Helena Hospital, St. Helena, California
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - NIH - Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Christian Hospital Northeast-Northwest, St Louis, Missouri
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mountainview Medical, Berlin Corners, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin

REFERENCES:
- [Derived] Morrison VA, Le-Rademacher J, Bobek O, Satele D, Leonard JP, Jatoi A. Association of age and performance status with adverse events in older adults with diffuse large B-cell lymphoma receiving frontline R-CHOP therapy: Alliance 151930, a secondary analysis of the phase III trial CALGB 50303. J Geriatr Oncol. 2025 Mar;16(2):102185. doi: 10.1016/j.jgo.2025.102185. Epub 2025 Jan 13. PMID 39809075
- [Derived] Schoder H, Polley MC, Knopp MV, Hall N, Kostakoglu L, Zhang J, Higley HR, Kelloff G, Liu H, Zelenetz AD, Cheson BD, Wagner-Johnston N, Kahl BS, Friedberg JW, Hsi ED, Leonard JP, Schwartz LH, Wilson WH, Bartlett NL. Prognostic value of interim FDG-PET in diffuse large cell lymphoma: results from the CALGB 50303 Clinical Trial. Blood. 2020 Jun 18;135(25):2224-2234. doi: 10.1182/blood.2019003277. PMID 32232481
- [Derived] Bartlett NL, Wilson WH, Jung SH, Hsi ED, Maurer MJ, Pederson LD, Polley MC, Pitcher BN, Cheson BD, Kahl BS, Friedberg JW, Staudt LM, Wagner-Johnston ND, Blum KA, Abramson JS, Reddy NM, Winter JN, Chang JE, Gopal AK, Chadburn A, Mathew S, Fisher RI, Richards KL, Schoder H, Zelenetz AD, Leonard JP. Dose-Adjusted EPOCH-R Compared With R-CHOP as Frontline Therapy for Diffuse Large B-Cell Lymphoma: Clinical Outcomes of the Phase III Intergroup Trial Alliance/CALGB 50303. J Clin Oncol. 2019 Jul 20;37(21):1790-1799. doi: 10.1200/JCO.18.01994. Epub 2019 Apr 2. PMID 30939090
- [Derived] Barta SK, Lee JY, Kaplan LD, Noy A, Sparano JA. Pooled analysis of AIDS malignancy consortium trials evaluating rituximab plus CHOP or infusional EPOCH chemotherapy in HIV-associated non-Hodgkin lymphoma. Cancer. 2012 Aug 15;118(16):3977-83. doi: 10.1002/cncr.26723. Epub 2011 Dec 16. PMID 22180164

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - R-CHOP: Patients receive the following treatment:>
  * Rituximab 375 mg/m^2 IV infusion on Day 1 prior to CHOP chemotherapy>
  * Cyclophosphamide 750 mg/m^2 IV on Day 1>
  * Doxorubicin 50 mg/m^2 IV on Day 1>
  * Vincristine 1.4 mg/m^2 IV (2 mg cap) on Day 1>
  * Prednisone 40 mg/m^2/day PO on Days 1-5>
  * filgrastim or pegfilgrastim as defined in the protocol> Required ancillary medications is administered during all cycles as defined in the protocol.> Cycles will be repeated every 21 days for 6 treatment cycles. Restaging will occur after Cycles 4 and 6.
- Arm B - DA-EPOCH-R: Patients receive the following treatment:> Cycle 1 Doses:>
  * Rituximab 375 mg/m^2 IV infusion on Day 1 prior to EPOCH chemotherapy>
  * Doxorubicin 10 mg/m^2/day CIVI on Days 1-4>
  * Etoposide 50 mg/m^2/day CIVI on Days 1-4>
  * Vincristine 0.4 mg/m^2/day (no cap) CIVI on Days 1-4 (total 1.6 mg/m2 over 96 hours)>
  * Cyclophosphamide 750 mg/m^2 IV on Day 5 (following completion of 96 hour infusions)>
  * Prednisone 60 mg/m^2 PO BID on Days 1-5>
  * Administer filgrastim 480 mcg subcutaneous daily from Day 6 until ANC > 5000 after the > nadir (nadir usually between Days 10-12) or for 10 days (Days 6-15) if the ANC is not > being monitored, during every cycle.> Doses for subsequent cycles will be determined by the absolute neutrophil (ANC) or platelet nadir from the previous cycle.> Required ancillary medications are administered during all cycles as defined in the protocol.> Cycles will be repeated every 21 days for a maximum of 6 cycles. Restaging will occur after Cycles 4 and 6.
Period: Overall Study
Arm/Group | Arm A - R-CHOP | Arm B - DA-EPOCH-R
Started | 262 | 262
Evaluable for Primary Endpoint | 250 | 241
Evaluable for Safety Analysis (Evaluable for adverse events) | 243 | 237
Completed | 250 | 241
Not Completed | 12 | 21

BASELINE CHARACTERISTICS:
Population: Participants who completed the study in the Participant Flow are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - R-CHOP | Arm B - DA-EPOCH-R | Total
Number analyzed (Participants) | 250 | 241 | 491
Age, Continuous [Median (Full Range); unit: years] — Population: Number analyzed in row differs from overall due to missing data.
  years
    number analyzed (Participants) | 247 | 239 | 486
    (all) | 58.0 [18.0 to 86.0] | 58.0 [19.0 to 84.0] | 58.0 [18.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall due to missing data.
  Participants
    number analyzed (Participants) | 249 | 241 | 490
    Female | 116 | 109 | 225
    Male | 133 | 132 | 265
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 31
  Not Hispanic or Latino | 220 | 214 | 434
  Unknown or Not Reported | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 29 | 31 | 60
  White | 196 | 189 | 385
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 11 | 8 | 19
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair. Population: The number analyzed in row differs from overall due to missing data.
  Participants
    number analyzed (Participants) | 249 | 241 | 490
    0 | 101 | 113 | 214
    1 | 119 | 96 | 215
    2 | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival Rate at 2 and 5 Years
Description: Progression-free survival (PFS) is defined as the time from randomization to progression, relapse, or death from any cause, whichever occurred first. Progression (PD) or Relapse>
  * ≥ 50% increase from nadir in the SPD of any previously identified abnormal node for PRs or nonresponders.>
  * Appearance of any new lesion during or after completion of therapy.>
  * PET+ is not a criterion for progressive disease. Patients only with PET+ findings must have evidence of progression on CT or biopsy proven.>
  The PFS rate (percentage of participants who are alive and progression-free) at 2 and 5 years Kaplan Meier estimates and 95% Confidence Intervals are reported below.
Time Frame: Up to 5 years post-registration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B - DA-EPOCH-R | Arm A - R-CHOP
Number analyzed (Participants) | 241 | 250
percentage of participants
  2-year PFS | 78.9 [73.8 to 84.2] | 75.5 [70.2 to 81.1]
  5-year PFS | 68.0 [62.1 to 74.5] | 66.0 [60.2 to 72.5]
Statistical Analysis 1: Comparison: Arm B - DA-EPOCH-R vs Arm A - R-CHOP; Test type: Superiority; p = 0.6519, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.68 to 1.27]

2. Secondary Outcome: Response Rate
Description: The overall response rate is defined as the percentage of participants with a response (Complete Response or Partial Response)
Time Frame: Up to 5 years post-registration
Measure: Number; unit: percentage of participants
Arm/Group | Arm B - DA-EPOCH-R | Arm A - R-CHOP
Number analyzed (Participants) | 241 | 250
percentage of participants | 86.7 | 88.0
Statistical Analysis 1: Comparison: Arm B - DA-EPOCH-R vs Arm A - R-CHOP; Test type: Superiority; p = 0.67, t-test, 2 sided

3. Secondary Outcome: Overall Survival Rate at 2 and 5 Years
Description: Overall survival is defined as the time from randomization to death due to any cause. The overall survival (OS) rate (percentage of participants who are still alive) at 2 and 5 years Kaplan Meier estimates and 95% confidence intervals are reported below.
Time Frame: Up to 5 years post-registration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm B - DA-EPOCH-R | Arm A - R-CHOP
Number analyzed (Participants) | 241 | 250
percentage of participants
  2-year OS rate | 86.5 [82.3 to 91.0] | 85.7 [81.4 to 90.2]
  5-year OS rate | 77.5 [72.2 to 83.2] | 78.5 [73.4 to 83.9]
Statistical Analysis 1: Comparison: Arm B - DA-EPOCH-R vs Arm A - R-CHOP; Test type: Superiority; p = 0.6414, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.75 to 1.59]

4. Other Pre Specified Outcome: Whether the Gene Expression Signatures That Were Previously Associated With Survival Following CHOP Therapy Are Associated With Survival in Either of the Treatment Arms of the Prospective Trial
Time Frame: Up to 5 years post-registration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: All participants are followed for survival (i.e. included in the All-cause mortality table). Participants who received at least one dose of treatment are evaluable for adverse events (i.e. included in the Serious AE and Other (Not Including Serious) AE tables).
Groups:
- Arm A - R-CHOP: Cycles will be repeated every 21 days for 6 treatment cycles. Restaging will occur after Cycles 4 and 6.
- Arm B - DA-EPOCH-R: Cycles will be repeated every 21 days for a maximum of 6 cycles. Restaging will occur after Cycles 4 and 6.
Arm/Group | Arm A - R-CHOP | Arm B - DA-EPOCH-R
All-Cause Mortality (participants affected / at risk) | 53/250 | 56/241
Serious Adverse Events (participants affected / at risk) | 232/243 | 214/237
Other Adverse Events (participants affected / at risk) | 94/243 | 119/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - R-CHOP (N=243) | Arm B - DA-EPOCH-R (N=237)
Febrile neutropenia (Blood and lymphatic system disorders) | 23 (26) | 43 (64)
Hemoglobin decreased (Blood and lymphatic system disorders) | 193 (488) | 201 (564)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (5)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 11 (17)
Anal mucositis (clin exam) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 84 (128) | 81 (119)
Diarrhea (Gastrointestinal disorders) | 13 (19) | 14 (14)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 4 (5)
Esophageal mucositis (clin exam) (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 3 (7)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 2 (2)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 13 (18) | 23 (28)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 18 (31) | 32 (55)
Nausea (Gastrointestinal disorders) | 21 (33) | 15 (25)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (9) | 7 (9)
Chest pain (General disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 2 (2) | 3 (3)
Death NOS (General disorders) | 3 (3) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 7 (9) | 9 (12)
Fatigue (General disorders) | 27 (41) | 41 (60)
Fever (General disorders) | 6 (6) | 2 (2)
Gait abnormal (General disorders) | 0 (0) | 1 (1)
General symptom (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2)
Sudden death (General disorders) | 0 (0) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 15 (18) | 9 (9)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 2 (3)
Bronchitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Colitis, infectious (Infections and infestations) | 0 (0) | 1 (1)
Device related infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Esophageal infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Esophageal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 3 (3)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 2 (4)
Nail infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Otitis media(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 0 (0)
Paranasal sinus infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 3 (4)
Pneumonia(unknown ANC) (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 1 (1)
Sepsis(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 2 (2)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 1 (1)
Tooth infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 1 (2)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 2 (3)
Vaginal infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Activated partial throm time prolonged (Investigations) | 1 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 5 (6) | 7 (10)
Alkaline phosphatase increased (Investigations) | 0 (0) | 6 (18)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 5 (6)
Blood bilirubin increased (Investigations) | 1 (1) | 4 (7)
CD4 lymphocytes decreased (Investigations) | 1 (4) | 2 (3)
Creatinine increased (Investigations) | 3 (6) | 5 (8)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 4 (7)
INR increased (Investigations) | 0 (0) | 1 (2)
Laboratory test abnormal (Investigations) | 2 (3) | 2 (2)
Leukocyte count decreased (Investigations) | 72 (117) | 105 (242)
Lymphocyte count decreased (Investigations) | 60 (114) | 86 (231)
Neutrophil count decreased (Investigations) | 179 (331) | 190 (506)
Platelet count decreased (Investigations) | 97 (182) | 184 (479)
Serum cholesterol increased (Investigations) | 1 (3) | 0 (0)
Weight loss (Investigations) | 4 (5) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (9) | 14 (17)
Blood glucose increased (Metabolism and nutrition disorders) | 20 (37) | 25 (39)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 22 (24) | 19 (22)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (4) | 12 (19)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (4) | 15 (28)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 5 (10)
Serum magnesium decreased (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 5 (11)
Serum phosphate decreased (Metabolism and nutrition disorders) | 5 (5) | 12 (14)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (6) | 29 (44)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 5 (5) | 6 (7)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 17 (28)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 5 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (5)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (4)
Arachnoiditis (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 10 (11) | 8 (10)
Dysgeusia (Nervous system disorders) | 4 (6) | 4 (7)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 14 (15)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 23 (31) | 36 (62)
Peripheral sensory neuropathy (Nervous system disorders) | 104 (186) | 141 (322)
Syncope (Nervous system disorders) | 2 (2) | 2 (2)
Tremor (Nervous system disorders) | 2 (2) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (4) | 5 (7)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 5 (8) | 7 (9)
Insomnia (Psychiatric disorders) | 8 (11) | 5 (6)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (2)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Testicular hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 9 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (funct/sympt) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (23) | 8 (19)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hand-and-foot syndrome/reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 9 (12)
Hypotension (Vascular disorders) | 0 (0) | 7 (11)
Thrombosis (Vascular disorders) | 6 (6) | 4 (5)
Vascular disorder (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - R-CHOP (N=243) | Arm B - DA-EPOCH-R (N=237)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 26 (27) | 44 (57)
Hemoglobin decreased (Blood and lymphatic system disorders) | 80 (126) | 116 (199)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 6 (7)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 6 (6) | 3 (3)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 7 (7)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 8 (9)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 18 (20) | 35 (45)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 14 (15)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 7 (7)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4) | 5 (6)
Jejunal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (clin exam) (Gastrointestinal disorders) | 3 (4) | 13 (19)
Mucositis oral (funct/sympt) (Gastrointestinal disorders) | 5 (5) | 17 (21)
Nausea (Gastrointestinal disorders) | 9 (9) | 13 (15)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 11 (12)
Chest pain (General disorders) | 1 (1) | 4 (4)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 10 (11) | 6 (6)
Fatigue (General disorders) | 14 (17) | 20 (23)
Fever (General disorders) | 3 (3) | 2 (2)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (3)
Visceral edema (General disorders) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 5 (5)
Immune system disorder (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal infection(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0)
Anorectal infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection(gr 0/1/2 ANC) (Infections and infestations) | 2 (2) | 1 (1)
Catheter related infection(gr 3/4 ANC) (Infections and infestations) | 4 (4) | 4 (4)
Colitis, infectious (Infections and infestations) | 1 (1) | 2 (3)
Esophageal infection(unknown ANC) (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 2 (2)
Infection(gr 0/1/2 ANC) (Infections and infestations) | 2 (3) | 6 (6)
Infectious colitis(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 2 (3)
Lip infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Lymph gland infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 2 (2)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0)
Pancreas infection(gr 3/4 ANC) (Infections and infestations) | 1 (1) | 0 (0)
Peritoneal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia(gr 0/1/2 ANC) (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia(gr 3/4 ANC) (Infections and infestations) | 4 (4) | 5 (5)
Pneumonia(unknown ANC) (Infections and infestations) | 1 (1) | 0 (0)
Sepsis(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Sepsis(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 3 (4)
Sepsis(unknown ANC) (Infections and infestations) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Skin infection(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 1 (1)
Tooth infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection(gr 3/4 ANC) (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory infectn(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection(gr 3/4 ANC) (Infections and infestations) | 3 (3) | 5 (6)
Vaginal infection(gr 0/1/2 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection(gr 3/4 ANC) (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection(gr 0/1/2 ANC) (Infections and infestations) | 1 (1) | 1 (1)
Wound infection(gr 3/4 ANC) (Infections and infestations) | 2 (2) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraop. inj. - Spinal cord (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Venous injury - Viscera (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial throm time prolonged (Investigations) | 0 (0) | 4 (4)
Alanine aminotransferase increased (Investigations) | 3 (3) | 6 (6)
Alkaline phosphatase increased (Investigations) | 2 (2) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 4 (4)
Blood bilirubin increased (Investigations) | 4 (4) | 4 (5)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 2 (3)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1)
Creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 3 (3)
Leukocyte count decreased (Investigations) | 42 (58) | 66 (106)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 34 (52) | 51 (93)
Neutrophil count decreased (Investigations) | 74 (109) | 107 (169)
Platelet count decreased (Investigations) | 53 (73) | 107 (167)
Serum cholesterol increased (Investigations) | 1 (1) | 4 (6)
Weight loss (Investigations) | 4 (4) | 4 (4)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 5 (6)
Blood glucose increased (Metabolism and nutrition disorders) | 12 (13) | 13 (18)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 16 (18) | 21 (28)
Serum albumin decreased (Metabolism and nutrition disorders) | 8 (10) | 19 (23)
Serum calcium decreased (Metabolism and nutrition disorders) | 7 (8) | 16 (20)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 5 (6) | 11 (14)
Serum potassium decreased (Metabolism and nutrition disorders) | 5 (5) | 23 (28)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (8) | 10 (13)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (10)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Mini mental status examination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5) | 16 (20)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (31) | 68 (108)
Seizure (Nervous system disorders) | 0 (0) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3) | 4 (4)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 9 (10)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (9)
Pharyngeal mucositis (clin exam) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 8 (8) | 13 (15)
Thrombosis (Vascular disorders) | 6 (6) | 10 (11)
Vascular disorder (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT00118209/Prot_SAP_000.pdf